CLINICAL TRIAL: NCT03255252
Title: Assessment Study to Evaluate Specific Immune Response in Locally Advanced Cervix Cancer After Radio-chemotherapy (IMMUVIX)
Brief Title: Assessment Study to Evaluate Specific Immune Response in Locally Advanced Cervix Cancer After Radio-chemotherapy
Acronym: IMMUVIX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC 2015/27
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: radiothérapy with concomittant chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cisplatin (Experimental): Weekly cisplatin (40 mg/m²) will be administered during radiotherapy. At least 3 cycles of cisplatin should be performed according to the hematological and renal functions but not mandatory.
  Interventions: Drug: Cisplatin injection; Combination Product: radiotherapy

INTERVENTIONS:
Drug: Cisplatin injection — Weekly cisplatin (40 mg/m²) will be administered during radiotherapy. At least 3 cycles of cisplatin should be performed according to the hematological and renal functions but not mandatory.
Combination Product: radiotherapy — A total dose of 45Gy in 25 fractions to the PTV is considered standard but simultaneous integrated boost or two steps boost to specific volumes (positive lymph nodes for example) are accepted and left to the investigator's discretion).

SUMMARY:
Perspectives:

* To set-up another clinical trial with this specific phenotype as the main stratification factor. Therefore a more aggressive or a more specific systemic treatment (with or without an immunomodulator) could be proposed to those selected patients in the field of personalized medicine.
* To evaluate the use of the smear as a surrogate non-invasive technique to biopsy for immunomonitoring.
* To use the CTC/PD-L1 assay as a liquid biopsy in future clinical trials for stratification and monitoring of cancer patients undergoing immune checkpoint treatments. This specific subset of CTCs might represent metastatic cells with a high potential to escape T cell-mediated lysis and might therefore be the actual targets of immunotherapy.

DETAILED DESCRIPTION:
Cervical cancer is a real worldwide health care issue. High-risk human papillomavirus (HR-HPV) chronic infection is a co-factor in the development of the cervical cancer.

The HR-HPV genome encodes two oncoproteins (E6 and E7) which are required to sustain the malignant phenotype of pre-neoplastic lesions and are considered as foreign antigens recognized by the immune system, Many studies have suggested that local immunologic escape can cause the emergence of HPV-induced cervical cancer Radio-chemotherapy is the gold standard treatment for locally advanced cervical cancer, resulting in 2 year-control rates of about 70 to 85 %. A better and earlier understanding of the reasons for tumor escape may hopefully help to improve these outcomes.

Both radiation and chemotherapy are myelosuppressive treatments, but new treatment modalities such as Intensity-Modulated Radiation Therapy (IMRT) may allow a more rapid hematologic recovery. In addition to this immunosuppressive microenvironment, a significant number of tumor-infiltrating lymphocytes (TILs) are detected in cervical cancer tissue, highlighting interactions between tumor and immune cells.

Another issue is the fact that cancer cells develop different strategies to bypass the immune surveillance, such as a down-regulation of class I human leucocyte antigen (HLA) on tumor cells surface.

Furthermore, there is growing evidence of the importance of immune cells in response to cervical cancer treatment. TILs have been correlated with cervical cancer patients' outcome. More precisely, the location and type of these immune cells seem to be of great importance for the tumor response to treatment.

Receptors with negative regulatory function have been identified on the surface of those T cells, including CTLA4 and PD1 and seem to play a great role in tumor escape to treatment.

The presence of circulating tumor cells (CTCs) was shown to be correlated with a poor patient's prognosis in many cancers. A recent study suggested a potential mechanism of immune escape of these CTCs resulting in metastasis spreading.

The hypothesis of this study is that the frequency of PD1+,CD39+, specific phenotype of the non-regulatory CD4+ and CD8+ T cells among TILs is involved with the lack of response to the treatment and correlates with an early relapse after the treatment (i.e. patients with a very poor prognosis).

Perspectives:

* To set-up another clinical trial with this specific phenotype as the main stratification factor. Therefore a more aggressive or a more specific systemic treatment (with or without an immunomodulator) could be proposed to those selected patients in the field of personalized medicine.
* To evaluate the use of the smear as a surrogate non-invasive technique to biopsy for immunomonitoring.
* To use the CTC/PD-L1 assay as a liquid biopsy in future clinical trials for stratification and monitoring of cancer patients undergoing immune checkpoint treatments. This specific subset of CTCs might represent metastatic cells with a high potential to escape T cell-mediated lysis and might therefore be the actual targets of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* HPV-positive cervical cancer proven* by biopsy.
* All FIGO stages cervical cancers which are the matter for radio-chemotherapy and exclusive brachytherapy indications.
* ECOG performance status ≤2.
* Ability to give informed consent.
* Patients must be affiliated to a Social Security System.
* Patient information and written informed consent form signed.

Exclusion Criteria:

* Adenocarcinoma of cervix.
* Known autoimmune disorder.
* History of HIV and/ or hepatitis infection.
* History of pelvic radiation or radio-chemotherapy.
* Recurrent or metastatic cervical cancer.
* Contra-indication for cisplatin.
* Patient pregnant and/or breastfeeding.
* History of other malignancy within the previous 5 years (except for appropriately treated melanoma skin carcinoma).
* Patients with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Expression of CD8+CD39+PD1+ lymphocytes infiltrate on cervix biopsies | through study completion, an average of 1 year disease free survival
  Cervix biopsies analysis

SECONDARY OUTCOMES:
Effect on 1-year DFS of other putative biomarkers (CD73, CD39, PD1 and Tim3) on the non-regulatory CD4+ and CD8+ lymphocytes | through study completion, an average of 1 year disease free survival
  Cervix biopsies and blood samples analysis

CONTACTS AND LOCATIONS:
Overall Officials: Riou Olivier, MD, Study Chair — ICM Val d'Aurelle
Locations (3):
- France (3):
  - Clinique Beausoleil, Montpellier
  - CHRU Montpellier, Montpellier
  - Moussin Aurore, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] De Vuyst H, Clifford G, Li N, Franceschi S. HPV infection in Europe. Eur J Cancer. 2009 Oct;45(15):2632-9. doi: 10.1016/j.ejca.2009.07.019. Epub 2009 Aug 24. PMID 19709878
- [Background] zur Hausen H. Papillomavirus infections--a major cause of human cancers. Biochim Biophys Acta. 1996 Oct 9;1288(2):F55-78. doi: 10.1016/0304-419x(96)00020-0. PMID 8876633
- [Background] Mauch P, Constine L, Greenberger J, Knospe W, Sullivan J, Liesveld JL, Deeg HJ. Hematopoietic stem cell compartment: acute and late effects of radiation therapy and chemotherapy. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1319-39. doi: 10.1016/0360-3016(94)00430-S. PMID 7713791
- [Background] Mell LK, Tiryaki H, Ahn KH, Mundt AJ, Roeske JC, Aydogan B. Dosimetric comparison of bone marrow-sparing intensity-modulated radiotherapy versus conventional techniques for treatment of cervical cancer. Int J Radiat Oncol Biol Phys. 2008 Aug 1;71(5):1504-10. doi: 10.1016/j.ijrobp.2008.04.046. PMID 18640499
- [Background] Kobayashi A, Weinberg V, Darragh T, Smith-McCune K. Evolving immunosuppressive microenvironment during human cervical carcinogenesis. Mucosal Immunol. 2008 Sep;1(5):412-20. doi: 10.1038/mi.2008.33. Epub 2008 Jul 2. PMID 19079205
- [Background] Jordanova ES, Gorter A, Ayachi O, Prins F, Durrant LG, Kenter GG, van der Burg SH, Fleuren GJ. Human leukocyte antigen class I, MHC class I chain-related molecule A, and CD8+/regulatory T-cell ratio: which variable determines survival of cervical cancer patients? Clin Cancer Res. 2008 Apr 1;14(7):2028-35. doi: 10.1158/1078-0432.CCR-07-4554. PMID 18381941
- [Background] Hasim A, Abudula M, Aimiduo R, Ma JQ, Jiao Z, Akula G, Wang T, Abudula A. Post-transcriptional and epigenetic regulation of antigen processing machinery (APM) components and HLA-I in cervical cancers from Uighur women. PLoS One. 2012;7(9):e44952. doi: 10.1371/journal.pone.0044952. Epub 2012 Sep 14. PMID 23024775
- [Background] Gadducci A, Guerrieri ME, Greco C. Tissue biomarkers as prognostic variables of cervical cancer. Crit Rev Oncol Hematol. 2013 May;86(2):104-29. doi: 10.1016/j.critrevonc.2012.09.003. Epub 2012 Sep 30. PMID 23031678
- [Background] Bell MC, Edwards RP, Partridge EE, Kuykendall K, Conner W, Gore H, Turbat-Herrara E, Crowley-Nowick PA. CD8+ T lymphocytes are recruited to neoplastic cervix. J Clin Immunol. 1995 May;15(3):130-6. doi: 10.1007/BF01543104. PMID 7559915
- [Background] Yamazawa K, Matsui H, Ishikura H, Seki K, Mitsuhashi A, Sekiya S. Significance of perivascular lymphocytic infiltrates on survival of patients with invasive cervical cancer. J Immunother. 2003 Mar-Apr;26(2):149-55. doi: 10.1097/00002371-200303000-00007. PMID 12616106
- [Background] Piersma SJ, Jordanova ES, van Poelgeest MI, Kwappenberg KM, van der Hulst JM, Drijfhout JW, Melief CJ, Kenter GG, Fleuren GJ, Offringa R, van der Burg SH. High number of intraepithelial CD8+ tumor-infiltrating lymphocytes is associated with the absence of lymph node metastases in patients with large early-stage cervical cancer. Cancer Res. 2007 Jan 1;67(1):354-61. doi: 10.1158/0008-5472.CAN-06-3388. PMID 17210718
- [Background] de Vos van Steenwijk PJ, Ramwadhdoebe TH, Goedemans R, Doorduijn EM, van Ham JJ, Gorter A, van Hall T, Kuijjer ML, van Poelgeest MI, van der Burg SH, Jordanova ES. Tumor-infiltrating CD14-positive myeloid cells and CD8-positive T-cells prolong survival in patients with cervical carcinoma. Int J Cancer. 2013 Dec 15;133(12):2884-94. doi: 10.1002/ijc.28309. Epub 2013 Jul 5. PMID 23740735
- [Background] Sznol M, Chen L. Antagonist antibodies to PD-1 and B7-H1 (PD-L1) in the treatment of advanced human cancer. Clin Cancer Res. 2013 Mar 1;19(5):1021-34. doi: 10.1158/1078-0432.CCR-12-2063. PMID 23460533
- [Background] Karim R, Jordanova ES, Piersma SJ, Kenter GG, Chen L, Boer JM, Melief CJ, van der Burg SH. Tumor-expressed B7-H1 and B7-DC in relation to PD-1+ T-cell infiltration and survival of patients with cervical carcinoma. Clin Cancer Res. 2009 Oct 15;15(20):6341-7. doi: 10.1158/1078-0432.CCR-09-1652. Epub 2009 Oct 13. PMID 19825956
- [Background] Yan J, Zhang Y, Zhang JP, Liang J, Li L, Zheng L. Tim-3 expression defines regulatory T cells in human tumors. PLoS One. 2013;8(3):e58006. doi: 10.1371/journal.pone.0058006. Epub 2013 Mar 5. PMID 23526963
- [Background] Bastid J, Cottalorda-Regairaz A, Alberici G, Bonnefoy N, Eliaou JF, Bensussan A. ENTPD1/CD39 is a promising therapeutic target in oncology. Oncogene. 2013 Apr 4;32(14):1743-51. doi: 10.1038/onc.2012.269. Epub 2012 Jul 2. PMID 22751118
- [Background] Bastid J, Regairaz A, Bonnefoy N, Dejou C, Giustiniani J, Laheurte C, Cochaud S, Laprevotte E, Funck-Brentano E, Hemon P, Gros L, Bec N, Larroque C, Alberici G, Bensussan A, Eliaou JF. Inhibition of CD39 enzymatic function at the surface of tumor cells alleviates their immunosuppressive activity. Cancer Immunol Res. 2015 Mar;3(3):254-65. doi: 10.1158/2326-6066.CIR-14-0018. Epub 2014 Nov 17. PMID 25403716
- [Background] Bonnefoy N, Bastid J, Alberici G, Bensussan A, Eliaou JF. CD39: A complementary target to immune checkpoints to counteract tumor-mediated immunosuppression. Oncoimmunology. 2015 Feb 3;4(5):e1003015. doi: 10.1080/2162402X.2014.1003015. eCollection 2015 May. PMID 26155397
- [Background] Ma Y, Adjemian S, Mattarollo SR, Yamazaki T, Aymeric L, Yang H, Portela Catani JP, Hannani D, Duret H, Steegh K, Martins I, Schlemmer F, Michaud M, Kepp O, Sukkurwala AQ, Menger L, Vacchelli E, Droin N, Galluzzi L, Krzysiek R, Gordon S, Taylor PR, Van Endert P, Solary E, Smyth MJ, Zitvogel L, Kroemer G. Anticancer chemotherapy-induced intratumoral recruitment and differentiation of antigen-presenting cells. Immunity. 2013 Apr 18;38(4):729-41. doi: 10.1016/j.immuni.2013.03.003. Epub 2013 Apr 4. PMID 23562161
- [Background] Ko A, Kanehisa A, Martins I, Senovilla L, Chargari C, Dugue D, Marino G, Kepp O, Michaud M, Perfettini JL, Kroemer G, Deutsch E. Autophagy inhibition radiosensitizes in vitro, yet reduces radioresponses in vivo due to deficient immunogenic signalling. Cell Death Differ. 2014 Jan;21(1):92-9. doi: 10.1038/cdd.2013.124. Epub 2013 Sep 13. PMID 24037090
- [Background] Evans EM, Man S, Evans AS, Borysiewicz LK. Infiltration of cervical cancer tissue with human papillomavirus-specific cytotoxic T-lymphocytes. Cancer Res. 1997 Jul 15;57(14):2943-50. PMID 9230206
- [Background] Hohn H, Pilch H, Gunzel S, Neukirch C, Freitag K, Necker A, Maeurer MJ. Human papillomavirus type 33 E7 peptides presented by HLA-DR*0402 to tumor-infiltrating T cells in cervical cancer. J Virol. 2000 Jul;74(14):6632-6. doi: 10.1128/jvi.74.14.6632-6636.2000. PMID 10864677
- [Background] Hohn H, Pilch H, Gunzel S, Neukirch C, Hilmes C, Kaufmann A, Seliger B, Maeurer MJ. CD4+ tumor-infiltrating lymphocytes in cervical cancer recognize HLA-DR-restricted peptides provided by human papillomavirus-E7. J Immunol. 1999 Nov 15;163(10):5715-22. PMID 10553103
- [Background] Hilders CG, Ras L, van Eendenburg JD, Nooyen Y, Fleuren GJ. Isolation and characterization of tumor-infiltrating lymphocytes from cervical carcinoma. Int J Cancer. 1994 Jun 15;57(6):805-13. doi: 10.1002/ijc.2910570608. PMID 8206676
- [Background] Santin AD, Bellone S, Palmieri M, Bossini B, Roman JJ, Cannon MJ, Bignotti E, Cane S, Pecorelli S. Induction of tumor-specific cytotoxicity in tumor infiltrating lymphocytes by HPV16 and HPV18 E7-pulsed autologous dendritic cells in patients with cancer of the uterine cervix. Gynecol Oncol. 2003 May;89(2):271-80. doi: 10.1016/s0090-8258(03)00083-0. PMID 12713991
- [Background] de Jong A, van Poelgeest MI, van der Hulst JM, Drijfhout JW, Fleuren GJ, Melief CJ, Kenter G, Offringa R, van der Burg SH. Human papillomavirus type 16-positive cervical cancer is associated with impaired CD4+ T-cell immunity against early antigens E2 and E6. Cancer Res. 2004 Aug 1;64(15):5449-55. doi: 10.1158/0008-5472.CAN-04-0831. PMID 15289354
- [Background] Kenter GG, Welters MJ, Valentijn AR, Lowik MJ, Berends-van der Meer DM, Vloon AP, Essahsah F, Fathers LM, Offringa R, Drijfhout JW, Wafelman AR, Oostendorp J, Fleuren GJ, van der Burg SH, Melief CJ. Vaccination against HPV-16 oncoproteins for vulvar intraepithelial neoplasia. N Engl J Med. 2009 Nov 5;361(19):1838-47. doi: 10.1056/NEJMoa0810097. PMID 19890126
- [Background] Heusinkveld M, Welters MJ, van Poelgeest MI, van der Hulst JM, Melief CJ, Fleuren GJ, Kenter GG, van der Burg SH. The detection of circulating human papillomavirus-specific T cells is associated with improved survival of patients with deeply infiltrating tumors. Int J Cancer. 2011 Jan 15;128(2):379-89. doi: 10.1002/ijc.25361. Epub 2010 Apr 5. PMID 20473854
- [Background] van der Burg SH, Ressing ME, Kwappenberg KM, de Jong A, Straathof K, de Jong J, Geluk A, van Meijgaarden KE, Franken KL, Ottenhoff TH, Fleuren GJ, Kenter G, Melief CJ, Offringa R. Natural T-helper immunity against human papillomavirus type 16 (HPV16) E7-derived peptide epitopes in patients with HPV16-positive cervical lesions: identification of 3 human leukocyte antigen class II-restricted epitopes. Int J Cancer. 2001 Mar 1;91(5):612-8. doi: 10.1002/1097-0215(200002)9999:99993.0.co;2-c. PMID 11267969
- [Background] Welters MJ, de Jong A, van den Eeden SJ, van der Hulst JM, Kwappenberg KM, Hassane S, Franken KL, Drijfhout JW, Fleuren GJ, Kenter G, Melief CJ, Offringa R, van der Burg SH. Frequent display of human papillomavirus type 16 E6-specific memory t-Helper cells in the healthy population as witness of previous viral encounter. Cancer Res. 2003 Feb 1;63(3):636-41. PMID 12566307
- [Background] Welters MJ, van der Logt P, van den Eeden SJ, Kwappenberg KM, Drijfhout JW, Fleuren GJ, Kenter GG, Melief CJ, van der Burg SH, Offringa R. Detection of human papillomavirus type 18 E6 and E7-specific CD4+ T-helper 1 immunity in relation to health versus disease. Int J Cancer. 2006 Feb 15;118(4):950-6. doi: 10.1002/ijc.21459. PMID 16152582
- [Background] Ressing ME, van Driel WJ, Celis E, Sette A, Brandt MP, Hartman M, Anholts JD, Schreuder GM, ter Harmsel WB, Fleuren GJ, Trimbos BJ, Kast WM, Melief CJ. Occasional memory cytotoxic T-cell responses of patients with human papillomavirus type 16-positive cervical lesions against a human leukocyte antigen-A *0201-restricted E7-encoded epitope. Cancer Res. 1996 Feb 1;56(3):582-8. PMID 8564975
- [Background] Bontkes HJ, de Gruijl TD, van den Muysenberg AJ, Verheijen RH, Stukart MJ, Meijer CJ, Scheper RJ, Stacey SN, Duggan-Keen MF, Stern PL, Man S, Borysiewicz LK, Walboomers JM. Human papillomavirus type 16 E6/E7-specific cytotoxic T lymphocytes in women with cervical neoplasia. Int J Cancer. 2000 Oct 1;88(1):92-8. PMID 10962445
- [Background] Luxton JC, Rowe AJ, Cridland JC, Coletart T, Wilson P, Shepherd PS. Proliferative T cell responses to the human papillomavirus type 16 E7 protein in women with cervical dysplasia and cervical carcinoma and in healthy individuals. J Gen Virol. 1996 Jul;77 ( Pt 7):1585-93. doi: 10.1099/0022-1317-77-7-1585. PMID 8758003
- [Background] Steinert G, Scholch S, Niemietz T, Iwata N, Garcia SA, Behrens B, Voigt A, Kloor M, Benner A, Bork U, Rahbari NN, Buchler MW, Stoecklein NH, Weitz J, Koch M. Immune escape and survival mechanisms in circulating tumor cells of colorectal cancer. Cancer Res. 2014 Mar 15;74(6):1694-704. doi: 10.1158/0008-5472.CAN-13-1885. Epub 2014 Mar 5. PMID 24599131
- [Background] Mazel M, Jacot W, Pantel K, Bartkowiak K, Topart D, Cayrefourcq L, Rossille D, Maudelonde T, Fest T, Alix-Panabieres C. Frequent expression of PD-L1 on circulating breast cancer cells. Mol Oncol. 2015 Nov;9(9):1773-82. doi: 10.1016/j.molonc.2015.05.009. Epub 2015 Jun 9. PMID 26093818
- [Background] Golden EB, Apetoh L. Radiotherapy and immunogenic cell death. Semin Radiat Oncol. 2015 Jan;25(1):11-7. doi: 10.1016/j.semradonc.2014.07.005. PMID 25481261
- [Background] Delgado FG, Martinez E, Cespedes MA, Bravo MM, Navas MC, Combita Rojas AL. Increase of human papillomavirus-16 E7-specific T helper type 1 response in peripheral blood of cervical cancer patients after radiotherapy. Immunology. 2009 Apr;126(4):523-34. doi: 10.1111/j.1365-2567.2008.02912.x. Epub 2008 Sep 5. PMID 18778290
- [Background] Lim K, Small W Jr, Portelance L, Creutzberg C, Jurgenliemk-Schulz IM, Mundt A, Mell LK, Mayr N, Viswanathan A, Jhingran A, Erickson B, De los Santos J, Gaffney D, Yashar C, Beriwal S, Wolfson A, Taylor A, Bosch W, El Naqa I, Fyles A; Gyn IMRT Consortium. Consensus guidelines for delineation of clinical target volume for intensity-modulated pelvic radiotherapy for the definitive treatment of cervix cancer. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):348-55. doi: 10.1016/j.ijrobp.2009.10.075. Epub 2010 May 14. PMID 20472347